CLINICAL TRIAL: NCT03675737
Title: A Phase 3, Randomized, Double-blind Clinical Study of Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy as First-line Treatment in Participants With HER2 Negative, Previously Untreated, Unresectable or Metastatic Gastric Orgastroesophageal Junction Adenocarcinoma (KEYNOTE-859)
Brief Title: Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy in Participants Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma (MK-3475-859/KEYNOTE-859)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-859; MK-3475-859 (Other: MSD); KEYNOTE-859 (Other: MSD); JAPIC-CTI (Registry Identifier: 194649); 2023-508890-10-00 (Registry Identifier: EU CT); U1111-1299-1405 (Registry Identifier: UTN); 2018-001757-27 (EudraCT Number)
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Stomach Neoplasms
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Fluorouracil; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Chemotherapy (FP or CAPOX regimen) (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 2 years) + physicians' choice of either cisplatin 80 mg/m^2 IV on Day 1 Q3W and 5-fluorouracil (5FU) 800 mg/m^2/day via continuous IV infusion on Days 1 to 5 Q3W (FP regimen) OR oxaliplatin 130 mg/m^2 IV on Day 1 Q3W + capecitabine 1000 mg/m^2 orally twice a day (BID) on Days 1 to 14 Q3W (CAPOX regimen).
  Participants who complete up to 35 administrations of pembrolizumab (approximately 2 years) or achieve a complete response (CR) but experience progression of disease (PD), can initiate a second course of pembrolizumab for up to 17 cycles (approximately 1 additional year).
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: 5-fluorouracil; Drug: oxaliplatin; Drug: capecitabine
- Placebo + Chemotherapy (FP or CAPOX regimen) (Active Comparator): Participants receive placebo on Day 1 Q3W for up to 35 cycles (approximately 2 years) + physicians' choice of either cisplatin 80 mg/m^2 IV on Day 1 Q3W and 5FU 800 mg/m^2/day via continuous IV infusion on Days 1 to 5 Q3W (FP regimen) OR oxaliplatin 130 mg/m^2 IV on Day 1 Q3W + capecitabine 1000 mg/m^2 orally BID on Days 1 to 14 Q3W (CAPOX regimen).
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil; Drug: oxaliplatin; Drug: capecitabine; Drug: Placebo for Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Administered as an IV infusion on Day 1 Q3W
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Chemotherapy (FP or CAPOX regimen)
Drug: Cisplatin — Administered as an IV infusion on Day 1 Q3W
  Other Names: PLATINOL®
Drug: 5-fluorouracil — Administered as a continuous IV infusion on Days 1-5 Q3W
  Other Names: ADRUCIL®; 5FU
Drug: oxaliplatin — Administered as an IV infusion on Day 1 Q3W
  Other Names: ELOXATIN®
Drug: capecitabine — Administered orally BID on Days 1 to 14 Q3W
  Other Names: XELODA®
Drug: Placebo for Pembrolizumab — Administered as an IV infusion on Day 1 Q3W
  Arms: Placebo + Chemotherapy (FP or CAPOX regimen)

SUMMARY:
The purpose of this study is to evaluate the efficacy of pembrolizumab (MK-3745) in combination with chemotherapy (Cisplatin combined with 5-Fluorouracil [FP regimen] or oxaliplatin combined with capecitabine [CAPOX regimen]) versus placebo in combination with chemotherapy (FP or CAPOX regimens) in the treatment of human epidermal growth factor receptor 2 (HER2) negative advanced gastric or GEJ adenocarcinoma in adult participants.

The primary hypotheses of this study are that pembrolizumab plus chemotherapy is superior to placebo plus chemotherapy in terms of overall survival (OS).

ELIGIBILITY:
Inclusion Criteria

* Has histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma with known programmed cell death ligand 1 (PD-L1) expression status
* Has human epidermal growth factor receptor 2 (HER2) negative cancer
* Male participants must agree to use contraception during the treatment period and through 95 days after the last dose of chemotherapy, refrain from donating sperm, and be abstinent from heterosexual intercourse, as their preferred and usual lifestyle, and agree to remain abstinent or must agree to use contraception per study protocol unless confirmed to be azoospermic during this period
* Female participants who are not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP) OR is a WOCBP who agrees to use contraception or be abstinent from heterosexual intercourse, as their preferred and usual lifestyle, during the treatment period and through 180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is last, and agrees not to donate eggs to others or freeze/store for her own use for the purpose of reproduction during this period
* Has measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator assessment
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Has provided tumor tissue sample deemed adequate for PD-L1 biomarker analysis
* Has provided tumor tissue sample for microsatellite instability (MSI) biomarker analysis
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 3 days prior to the start of study intervention
* Has adequate organ function as demonstrated by laboratory testing within 10 days prior to the start of study treatment

Exclusion Criteria

* Has squamous cell or undifferentiated gastric cancer
* Has had major surgery, open biopsy, or significant traumatic injury within 28 days prior to randomization, anticipation of the need for major surgery during the course of study intervention, or has not recovered adequately from the toxicity and/or complications from previous surgery
* Has preexisting peripheral neuropathy >Grade 1
* Is a WOCBP who has a positive urine pregnancy test within 24 hours for urine or within 72 hours for serum prior to randomization or treatment allocation
* Has had previous therapy for locally advanced, unresectable or metastatic gastric/GEJ cancer. Participants may have received prior neoadjuvant and/or adjuvant therapy as long as it was completed ≥6 months prior to randomization
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1 or anti-programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX- 40, CD137)
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks prior to randomization or has not recovered from all adverse events (AEs) due to any previous therapies to ≤Grade 1 or baseline
* Has received prior radiotherapy within 2 weeks prior to study start or has not recovered from all previous radiation-related toxicities, required corticosteroids, and have not had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy
* Has known active CNS metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as Hepatitis C virus [HCV] ribonucleic acid [RNA] detected qualitatively) infection
* Has a known history of active tuberculosis
* Has hypokalemia (serum potassium less than the lower limit of normal)
* Has hypomagnesemia (serum magnesium less than the lower limit of normal)
* Has hypocalcemia (serum calcium less than the lower limit of normal)
* Has a history or current evidence of any condition (eg, known deficiency of the enzyme dihydropyrimidine dehydrogenase), therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is last
* Has had an allogenic tissue/solid organ transplant
* Has a known severe hypersensitivity (≥ Grade 3) to any of the study chemotherapy agents (including, but not limited to, infusional 5-fluorouracil or oral capecitabine) and/or to any of their excipients
* For participants taking cisplatin: has Grade ≥2 audiometric hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1579 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2025-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (215):
- United States (10):
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 120) ( Site 0124), Los Angeles, California
  - UC Irvine Health/Division of Hematology Oncology, Dept of Medicine ( Site 0128), Orange, California
  - University of Miami, Sylvester Comprehensive Cancer Center ( Site 0113), Miami, Florida
  - Greater Baltimore Medical Center ( Site 0102), Baltimore, Maryland
  - Minnesota Oncology Hematology, PA ( Site 8000), Minneapolis, Minnesota
  - University of Rochester ( Site 0122), Rochester, New York
  - Cancer Treatment Centers of America - Philadelphia ( Site 0112), Philadelphia, Pennsylvania
  - Allegheny General Hospital ( Site 0118), Pittsburgh, Pennsylvania
  - Oncology & Hematology Assoc. SW Virginia, Inc., DBA Blue Ridge Cancer Care ( Site 8001), Roanoke, Virginia
  - Wenatchee Valley Clinic [Wenatchee, WA] ( Site 0116), Wenatchee, Washington
- Argentina (5):
  - Instituto Medico Alexander Fleming ( Site 0307), Buenos Aires, Buenos Aires F.D.
  - Instituto de Investigaciones Metabolicas ( Site 0312), Buenos Aires
  - Fundacion Favaloro - Hospital Universitario ( Site 0302), Buenos Aires
  - Centro Oncologico Riojano Integral ( Site 0313), La Rioja
  - Instituto San Marcos ( Site 0311), San Juan
- Australia (3):
  - Liverpool Hospital ( Site 2301), Liverpool, New South Wales
  - Southern Medical Day Care Centre ( Site 2303), Wollongong, New South Wales
  - Box Hill Hospital ( Site 2300), Box Hill, Victoria
- Brazil (7):
  - Instituto do Cancer do Ceara ( Site 0407), Fortaleza, Ceará
  - CIONC - Centro Integrado de Oncologia de Curitiba ( Site 0405), Curitiba, Paraná
  - Hospital de Caridade de Ijui ( Site 0402), Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao ( Site 0403), Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncologicas ( Site 0400), Florianópolis, Santa Catarina
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0401), Rio de Janeiro
  - IBCC - Instituto Brasileiro de Controle do Cancer ( Site 0404), São Paulo
- Canada (4):
  - BC Cancer - Abbotsford ( Site 0206), Abbotsford, British Columbia
  - Sunnybrook Research Institute ( Site 0202), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0203), Toronto, Ontario
  - McGill University Health Centre ( Site 0208), Montreal, Quebec
- Chile (4):
  - Fundacion Arturo Lopez Perez FALP ( Site 0501), Santiago, Region M. de Santiago
  - Sociedad Oncovida S.A. ( Site 0508), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0502), Santiago, Region M. de Santiago
  - Instituto Clinico Oncologico del Sur ( Site 0500), Temuco, Región de la Araucanía
- China (29):
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 2421), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 2425), Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital ( Site 2410), Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital ( Site 2414), Fuzhou, Fujian
  - 900 Hospital of the Joint ( Site 2418), Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 2430), Xiamen, Fujian
  - Zhongshan Hospital Xiamen University ( Site 2447), Xiamen, Fujian
  - Guangdong General Hospital ( Site 2431), Guangzhou, Guangdong
  - Peking University Shenzhen Hospital ( Site 2442), Shenzhen, Guangdong
  - Fourth Hospital Of Hebei Medical University ( Site 2436), Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital ( Site 2401), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2415), Zhengzhou, Henan
  - Hubei Cancer Hospital ( Site 2434), Wuhan, Hubei
  - Xiangya Hospital Central-South University ( Site 2419), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 2439), Changsha, Hunan
  - Changzhou Cancer Hospital-Changzhou Fourth Peoples Hospital ( Site 2441), Changzhou, Jiangsu
  - The 81st Hospital of PLA ( Site 2413), Nanjing, Jiangsu
  - Jiangsu Cancer Hospital ( Site 2432), Nanjing, Jiangsu
  - Yancheng First People s Hospital ( Site 2426), Yancheng, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 2440), Nanchang, Jiangxi
  - The First Hospital of Jilin University ( Site 2416), Changchun, Jilin
  - The Affiliated Hospital of Qingdao University ( Site 2405), Qingdao, Shandong
  - Shanghai East Hospital ( Site 2403), Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University ( Site 2407), Shanghai, Shanghai Municipality
  - 1st Affil hosp of Med College of Xi'an Jiaotong University ( Site 2428), XiAn, Shanxi
  - Cancer Hospital Affiliated to Xinjiang Medical University ( Site 2420), Ürümqi, Xinjiang
  - Zhejiang Provincial People's Hospital ( Site 2446), Hangzhou, Zhejiang
  - Sir Run Run Show Hospital ( Site 2427), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2417), Hangzhou, Zhejiang
- Colombia (4):
  - Instituto Nacional de Cancerologia E.S.E ( Site 0605), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0608), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 0606), Montería, Departamento de Córdoba
  - Centro Medico Imbanaco de Cali S.A ( Site 0604), Cali, Valle del Cauca Department
- Costa Rica (3):
  - CIMCA Centro de Investigacion y Manejo del Cancer ( Site 3001), San José
  - Policlinico San Bosco ( Site 3002), San José
  - ICIMED - Instituto de Investigacion en Ciencias Medicas ( Site 3000), San José
- Czechia (6):
  - FN Ostrava ( Site 3105), Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice Plzen ( Site 3102), Pilsen, Plzeň Region
  - Masarykuv onkologicky ustav ( Site 3103), Brno, South Moravian
  - Nemocnice AGEL Novy Jicin a.s. ( Site 3104), Nový Jičín
  - Fakultni nemocnice Olomouc ( Site 3100), Olomouc
  - Fakultni Thomayerova nemocnice ( Site 3101), Prague
- Denmark (3):
  - Rigshospitalet ( Site 3202), Copenhagen, Capital Region
  - Aalborg University Hospital ( Site 3204), Aalborg, North Denmark
  - Odense Universitets Hospital ( Site 3201), Odense, Region Syddanmark
- France (7):
  - CHU de Rouen ( Site 1006), Rouen, Ain
  - CHU-Jean Minjoz ( Site 1002), Besançon, Doubs
  - C.H.R.U. de Brest - Hopital Morvan ( Site 1007), Brest, Finistere
  - Centre Oscar Lambret ( Site 1003), Lille, Nord
  - Institut de Cancerologie de l Ouest Centre Rene Gauducheau ( Site 1004), Saint-Herblain, Val-de-Marne
  - Institut Gustave Roussy ( Site 1000), Villejuif, Val-de-Marne
  - CHU Hopital Saint Antoine ( Site 1001), Paris
- Germany (5):
  - SLK-Kliniken Heilbronn ( Site 1104), Heilbronn, Baden-Wurttemberg
  - Universitaetsklinikum Leipzig ( Site 1114), Leipzig, Saxony
  - Charite Universitaetsmedizin Berlin ( Site 1101), Berlin
  - Facharztzentrum Eppendorf ( Site 1121), Hamburg
  - Asklepios Klinik Altona ( Site 1100), Hamburg
- Guatemala (5):
  - Celan SA ( Site 0705), Guatemala City
  - Oncomedica ( Site 0702), Guatemala City
  - Grupo Angeles SA ( Site 0701), Guatemala City
  - MEDI-K CAYALA ( Site 0704), Guatemala City
  - Centro Regional de Sub Especialidades Medicas SA ( Site 0703), Quetzaltenango
- Hong Kong (3):
  - Prince of Wales Hospital ( Site 2503), Hong Kong
  - Princess Margaret Hospital. ( Site 2502), Hong Kong
  - Queen Mary Hospital ( Site 2501), Hong Kong
- Hungary (5):
  - Bacs-Kiskun Megyei Korhaz ( Site 3306), Kecskemét, Bács-Kiskun county
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Gyula Korhaz-Rendelointezet ( Site 3302), Szolnok, Jász-Nagykun-Szolnok
  - Semmelweis Egyetem.. ( Site 3305), Budapest
  - Orszagos Onkologiai Intezet ( Site 3303), Budapest
  - University of Debrecen Medical Center Clinic of Oncology ( Site 3300), Debrecen
- Ireland (3):
  - St. James s Hospital ( Site 1200), Dublin
  - Beaumont Hospital ( Site 2101), Dublin
  - Tallaght University Hospital ( Site 1202), Dublin
- Israel (8):
  - Hadassah Ein Karem Jerusalem ( Site 1301), Jerusalem, Jerusalem
  - Chaim Sheba Medical Center ( Site 1304), Ramat Gan, Tel Aviv
  - Edith Wolfson Medical Center ( Site 1307), Holon, Tell Abib
  - Sourasky Medical Center ( Site 1306), Tel Aviv, Tell Abib
  - Soroka University Medical Center ( Site 1305), Beersheba
  - Rambam Medical Center ( Site 1303), Haifa
  - Meir Medical Center ( Site 1308), Kfar Saba
  - Rabin Medical Center ( Site 1302), Petah Tikva
- Italy (4):
  - Istituto Europeo di Oncologia ( Site 1411), Milan, Lombardy
  - Istituto Nazionale dei Tumori Fondazione IRCSS ( Site 1402), Milan
  - Istituto Oncologico Veneto ( Site 1412), Padua
  - Azienda Ospedaliera San Camillo Forlanini ( Site 1413), Roma
- Japan (20):
  - Aichi Cancer Center Hospital ( Site 2619), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2617), Kashiwa, Chiba
  - Hyogo Cancer Center ( Site 2604), Akashi, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 2603), Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 2610), Kasama, Ibaraki
  - Kagawa University Hospital ( Site 2615), Kita-gun, Kagawa-ken
  - Kitasato University Hospital ( Site 2618), Sagamihara, Kanagawa
  - Kanagawa Cancer Center ( Site 2614), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 2608), Hirakata, Osaka
  - Kindai University Hospital ( Site 2616), Sayama, Osaka
  - Osaka University Hospital ( Site 2600), Suita, Osaka
  - Saitama Cancer Center ( Site 2601), Kitaadachi-gun, Saitama
  - National Hospital Organization Kyushu Cancer Center ( Site 2612), Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2611), Hiroshima
  - Kumamoto University Hospital ( Site 2602), Kumamoto
  - Niigata Cancer Center Hospital ( Site 2613), Niigata
  - Osaka International Cancer Institute ( Site 2607), Osaka
  - National Cancer Center Hospital ( Site 2606), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 2605), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 2609), Tokyo
- Mexico (5):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0808), Guadalajara, Jalisco
  - Christus Muguerza Clinica Vidriera ( Site 0802), Monterrey, Nuevo León
  - Instituto Nacional de Cancerologia. ( Site 0804), Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0806), Mexico City
  - Medical Care and Research S.A. de C.V. ( Site 0809), Mérida
- Auckland City Hospital ( Site 2700), Auckland, Northland, New Zealand
- Peru (4):
  - Clinica Ricardo Palma Instituto de Oncologia y Radioterapia ( Site 0908), Lima
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 0901), Lima
  - Hospital Nacional Arzobispo Loayza ( Site 0902), Lima
  - Clinica San Gabriel ( Site 0907), Lima
- Poland (7):
  - Przychodnia Lekarska Komed ( Site 1514), Konin, Greater Poland Voivodeship
  - Szpital Uniwersytecki w Krakowie ( Site 1503), Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego ( Site 1506), Wroclaw, Lower Silesian Voivodeship
  - Dolnoslaskie Centrum Onkologii we Wroclawiu ( Site 1504), Wroclaw, Lower Silesian Voivodeship
  - Magodent Szpital Elblaska ( Site 1509), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Regionalny Szpital Specjalistyczny im Wl. Bieganskiego w Grudziadzu ( Site 1505), Grudziądz
- Russia (6):
  - Chelyabinsk Regional Clinical Oncology Dispensary-Chemotherapy ( Site 1608), Chelyabinsk, Chelyabinsk Oblast
  - SBHI Leningrad Regional Clinical Hospital ( Site 1616), Saint Petersburg, Leningradskaya Oblast'
  - Blokhin National Medical Oncology ( Site 1604), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 1614), Moscow, Moscow
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 1609), Samara, Samara Oblast
  - City Clinical Oncology Center ( Site 1603), Saint Petersburg, Sankt-Peterburg
- South Africa (10):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 1708), Port Elizabeth, Eastern Cape
  - Universitas Annex National Hospital ( Site 1701), Bloemfontein, Free State
  - Sandton Oncology Medical Group PTY LTD ( Site 1700), Johannesburg, Gauteng
  - Wits Clinical Research ( Site 1707), Parktown-Johannesburg, Gauteng
  - Tshwane District Hospital ( Site 1702), Pretoria, Gauteng
  - The Oncology Centre Overport and Umhlanga ( Site 1705), Durban, KwaZulu-Natal
  - Cancercare Rondebosch Oncology ( Site 1709), Cape Town, Western Cape
  - Groote Schuur Hospital ( Site 1706), Cape Town, Western Cape
  - Outeniqua Cancercare Oncology Unit ( Site 1704), George, Western Cape
  - Cape Town Oncology Trials Pty Ltd ( Site 1703), Kraaifontein, Western Cape
- South Korea (4):
  - Seoul National University Hospital ( Site 2803), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2800), Seoul
  - Asan Medical Center ( Site 2802), Seoul
  - Samsung Medical Center ( Site 2801), Seoul
- Spain (6):
  - Hospital General Universitario de Elche ( Site 1803), Elche, Alicante
  - Institut Catala d Oncologia Hospital Germans Trias i Pujol ( Site 1806), Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla ( Site 1804), Santander, Cantabria
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 1805), Pozuelo de Alarcón, Madrid
  - Hospital Universitario General de Asturias ( Site 1802), Oviedo, Principality of Asturias
  - Hospital General Universitari Vall d Hebron ( Site 1801), Barcelona
- Switzerland (7):
  - Universitaetsspital Basel ( Site 1900), Basel, Canton of Basel-City
  - Hopitaux Universitaires de Geneve HUG ( Site 1907), Geneva, Canton of Geneva
  - Kantonsspital St. Gallen ( Site 1901), Sankt Gallen, Canton of St. Gallen
  - Universitaetsspital Zuerich ( Site 1902), Zurich, Canton of Zurich
  - Istituto Oncologica della Svizzera Italiana (IOSI) ( Site 1905), Bellinzona, Canton Ticino
  - Kantonsspital Graubuenden ( Site 1903), Chur, Kanton Graubünden
  - Luzern Kantonsspital ( Site 1904), Lucerne
- Taiwan (4):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 2902), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 2901), Tainan
  - National Taiwan University Hospital ( Site 2900), Taipei
  - Mackay Memorial Hospital ( Site 2903), Taipei
- Turkey (Türkiye) (9):
  - Adana Sehir Hastanesi ( Site 2002), Adana
  - Hacettepe University Medical Faculty ( Site 2017), Ankara
  - Abdurrahman Yurtaslan Onkoloji Egitim ve Arastirma Hastanesi ( Site 2006), Ankara
  - Trakya Universitesi Tip Fakultesi ( Site 2015), Edirne
  - Ataturk Universitesi Tip Fakultesi Hastanesi ( Site 2000), Erzurum
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 2001), Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi ( Site 2011), Izmir
  - Malatya Inonu Universitesi Tip Fakultesi Hastanesi ( Site 2009), Malatya
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi ( Site 2012), Sakarya
- Ukraine (10):
  - City Clinical Hosp.4 of DCC ( Site 2201), Dnipro, Dnipropetrovsk Oblast
  - MI Kryviy Rih Center of Dnipropetrovsk Regional Council ( Site 2200), Kryviy Rih, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 2204), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 2208), Kharkiv, Kharkivs’ka Oblast’
  - Clinic of National Cancer Institute ( Site 2203), Kyiv, Kyivska Oblast
  - Medical and Diagnostic Centre LLC Dobryi Prognoz ( Site 2205), Kyiv, Kyivska Oblast
  - Lviv State Oncology Regional Treatment and Diagnostic Center ( Site 2210), Lviv, Lviv Oblast
  - MI Odessa Regional Oncological Centre ( Site 2212), Odesa, Odesa Oblast
  - Medical Centre LLC Oncolife ( Site 2202), Zaporizhzhya, Zaporizhzhia Oblast
  - Kyiv City Clinical Oncology Centre ( Site 2213), Kyiv
- United Kingdom (4):
  - South Devon Healthcare Foundation Trust. Torbay Hospital ( Site 1205), Torquay, Devon
  - Castle Hill Hospital ( Site 1201), Cottingham, East Riding Of Yorkshire
  - University College London Hospital ( Site 1211), London, London, City of
  - St. Georges University Hospital NHS Foundation Trust ( Site 1204), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Rha SY, Oh DY, Yanez P, Bai Y, Ryu MH, Lee J, Rivera F, Alves GV, Garrido M, Shiu KK, Fernandez MG, Li J, Lowery MA, Cil T, Cruz FM, Qin S, Luo S, Pan H, Wainberg ZA, Yin L, Bordia S, Bhagia P, Wyrwicz LS; KEYNOTE-859 investigators. Pembrolizumab plus chemotherapy versus placebo plus chemotherapy for HER2-negative advanced gastric cancer (KEYNOTE-859): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2023 Nov;24(11):1181-1195. doi: 10.1016/S1470-2045(23)00515-6. Epub 2023 Oct 21. PMID 37875143
- [Result] Qin S, Bai Y, Li J, Pan H, Luo S, Qu Y, Ye F, Yang L, Liu T, Li W, Chen X, Yang J, Ying J, Lin X, Zhao L, Liang X, Mao Y, Guo R, Zuo Y, Bordia S, Li S. First-Line Pembrolizumab Plus Chemotherapy for HER2-Negative Advanced Gastric Cancer: China Subgroup Analysis of the Randomized Phase 3 KEYNOTE-859 Study. Adv Ther. 2025 Apr;42(4):1892-1906. doi: 10.1007/s12325-024-03069-4. Epub 2025 Mar 1. PMID 40025394
- [Derived] Yasui H, Aizawa M, Yamaguchi K, Kawazoe A, Hara H, Tsuda M, Shoji H, Sugimoto N, Shibata N, Amagai K, Choda Y, Iwagami S, Esaki T, Kadowaki S, Shiratori S, Han S, Bordia S, Shitara K. First-line pembrolizumab plus chemotherapy for participants in Japan with gastric or gastroesophageal junction adenocarcinoma: subgroup analysis of the phase 3 KEYNOTE-859 study. Int J Clin Oncol. 2025 Oct;30(10):2003-2011. doi: 10.1007/s10147-025-02847-6. Epub 2025 Aug 1. PMID 40750941
- [Derived] Tabernero J, Bang YJ, Van Cutsem E, Fuchs CS, Janjigian YY, Bhagia P, Li K, Adelberg D, Qin SK. KEYNOTE-859: a Phase III study of pembrolizumab plus chemotherapy in gastric/gastroesophageal junction adenocarcinoma. Future Oncol. 2021 Aug;17(22):2847-2855. doi: 10.2217/fon-2021-0176. Epub 2021 May 12. PMID 33975465
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26343&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Chemotherapy (FP or CAPOX Regimen): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 2 years) + physicians' choice of either cisplatin 80 mg/m^2 IV on Day 1 Q3W and 5-fluorouracil (5FU) 800 mg/m^2/day via continuous IV infusion on Days 1 to 5 Q3W (FP regimen) OR oxaliplatin 130 mg/m^2 IV on Day 1 Q3W + capecitabine 1000 mg/m^2 orally twice a day (BID) on Days 1 to 14 Q3W (CAPOX regimen).
  Participants who completed up to 35 administrations of pembrolizumab (approximately 2 years) or achieved a complete response (CR) but experienced progression of disease (PD), could have initiated a second course of pembrolizumab for up to 17 cycles (approximately 1 additional year).
- Placebo + Chemotherapy (FP or CAPOX Regimen): Participants received placebo on Day 1 Q3W for up to 35 cycles (approximately 2 years) + physicians' choice of either cisplatin 80 mg/m^2 IV on Day 1 Q3W and 5FU 800 mg/m^2/day via continuous IV infusion on Days 1 to 5 Q3W (FP regimen) OR oxaliplatin 130 mg/m^2 IV on Day 1 Q3W + capecitabine 1000 mg/m^2 orally BID on Days 1 to 14 Q3W (CAPOX regimen).
Period: Overall Study
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Started | 790 | 789
Treated | 785 | 787
Completed | 0 | 0
Not Completed | 790 | 789
Not completed — Death | 593 | 660
Not completed — Lost to Follow-up | 1 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 14 | 12
Not completed — Ongoing in Study | 181 | 112

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen) | Total
Number analyzed (Participants) | 790 | 789 | 1579
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (11.9) | 60.0 (11.8) | 59.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 245 | 508
  Male | 527 | 544 | 1071
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 175 | 157 | 332
  Not Hispanic or Latino | 590 | 615 | 1205
  Unknown or Not Reported | 25 | 17 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 31 | 36 | 67
  Asian | 270 | 269 | 539
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 12 | 9 | 21
  White | 426 | 435 | 861
  More than one race | 43 | 30 | 73
  Unknown or Not Reported | 7 | 8 | 15
Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) <1 and CPS ≥1 Status [Count of Participants; unit: Participants] — PD-L1 positivity at baseline was determined by immunohistochemistry (IHC) using both tumor and blood cells. Participants were stratified (CPS <1 versus CPS ≥1) and some efficacy outcome measures were presented using a CPS cutoff of CPS ≥1 at baseline. Participants with a CPS <1 were classified as PD-L1 negative, participants with a CPS≥1 were classified as PD-L1 positive.
  Participants
    CPS ≥1 | 618 | 617 | 1235
    CPS <1 | 172 | 172 | 344
Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10 Status [Count of Participants; unit: Participants] — PD-L1 positivity at baseline was determined by immunohistochemistry (IHC) using both tumor and blood cells. Some efficacy outcome measures were presented using a CPS cutoff of CPS ≥10 at baseline. Participants with a CPS ≥10 were classified as PD-L1 strongly positive.
  Participants
    CPS ≥10 | 279 | 272 | 551
    CPS <10 | 509 | 517 | 1026
    Unknown | 2 | 0 | 2
Chemotherapy Regimen [Count of Participants; unit: Participants] — Participants received the physicians' choice of either the FP chemotherapy regimen (cisplatin and 5FU) OR the CAPOX regimen (oxaliplatin and capecitabine). Participants were stratified by chemotherapy regimen.
  Participants
    FP Regimen | 108 | 108 | 216
    CAPOX Regimen | 682 | 681 | 1363
Geographic Region [Count of Participants; unit: Participants] — Participants were stratified by geographic region using the following categories: Western Europe/Israel/North America/Australia; Asia; and Rest of World.
  Participants
    Western Europe/Israel/North America/Australia | 201 | 202 | 403
    Asia | 263 | 262 | 525
    Rest of World | 326 | 325 | 651

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in All Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. OS was estimated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to 45.9 months
Population: The analysis population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 790 | 789
Months | 12.9 [11.9 to 14.0] | 11.5 [10.6 to 12.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p < 0.0001, Log Rank — One-sided p-value based on log-rank test stratified by geographic region, Programmed Cell Death Ligand 1 (PD-L1) status (Combined Positive Score [CPS] <1 versus CPS ≥1), and chemotherapy regimen with small strata collapsed; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.70 to 0.87] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region, PD-L1 status (CPS <1 versus CPS ≥1), and chemotherapy regimen with small strata collapsed

2. Primary Outcome: Overall Survival (OS) In Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1
Description: as for outcome 1
Time Frame: Up to 45.9 months
Population: The analysis population included randomized participants with a PD-L1 CPS of ≥1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 618 | 617
Months | 13.0 [11.6 to 14.2] | 11.4 [10.5 to 12.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p < 0.0001, Log Rank — One-sided p-value based on log-rank test stratified by geographic region and chemotherapy regimen with small strata collapsed; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.65 to 0.84] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region and chemotherapy regimen with small strata collapsed

3. Primary Outcome: Overall Survival (OS) In Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10
Description: as for outcome 1
Time Frame: Up to 45.9 months
Population: The analysis population included randomized participants with a PD-L1 CPS of ≥10.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 279 | 272
Months | 15.7 [13.8 to 19.3] | 11.8 [10.3 to 12.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.53 to 0.79] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in All Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1 as assessed by BICR, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. PFS was estimated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to 49.5 months
Population: The analysis population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 790 | 789
Months | 6.9 [6.3 to 7.2] | 5.6 [5.5 to 5.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.67 to 0.85] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1
Description: as for outcome 4
Time Frame: Up to 49.5 months
Population: The analysis population included randomized participants with a PD-L1 CPS ≥1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 618 | 617
Months | 6.9 [6.0 to 7.2] | 5.6 [5.4 to 5.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.63 to 0.82] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10
Description: as for outcome 4
Time Frame: Up to 49.5 months
Population: The analysis population included randomized participants with a PD-L1 CPS ≥10.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 279 | 272
Months | 8.1 [6.8 to 8.5] | 5.6 [5.4 to 6.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.51 to 0.76] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in All Participants
Description: ORR was defined as the percentage of the participants who had a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 as assessed by BICR.
Time Frame: Up to 49.5 months
Population: The analysis population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 790 | 789
Percentage of Participants | 51.3 [47.7 to 54.8] | 42.0 [38.5 to 45.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p = 0.00009, Miettinen & Nurminen method — One-sided p-value based on Miettinen & Nurminen method stratified by geographic region, Programmed Cell Death Ligand 1 (PD-L1) status (Combined Positive Score [CPS] <1 versus CPS ≥1), and chemotherapy regimen with small strata collapsed; Difference in Percentage = 9.3, 95% CI 2-sided [4.4 to 14.1] — Based on Miettinen & Nurminen method stratified by geographic region, PD-L1 status (CPS <1 versus CPS ≥1), and chemotherapy regimen with small strata collapsed

8. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1
Description: as for outcome 7
Time Frame: Up to 49.5 months
Population: The analysis population included randomized participants with a PD-L1 CPS ≥1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 618 | 617
Percentage of Participants | 52.1 [48.1 to 56.1] | 42.6 [38.7 to 46.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p = 0.00041, Miettinen & Nurminen method — One-sided p-value based on Miettinen & Nurminen method stratified by geographic region and chemotherapy regimen with small strata collapsed; Difference in Percentage = 9.5, 95% CI 2-sided [3.9 to 15.0] — Based on Miettinen & Nurminen method stratified by geographic region and chemotherapy regimen with small strata collapsed

9. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10
Description: as for outcome 7
Time Frame: Up to 49.5 months
Population: The analysis population included randomized participants with a PD-L1 CPS ≥10.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 279 | 272
Percentage of Participants | 60.6 [54.6 to 66.3] | 43.0 [37.1 to 49.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) vs Placebo + Chemotherapy (FP or CAPOX Regimen); Test type: Superiority; p = 0.00002, Miettinen & Nurminen method — [p-value comment as in outcome 8, analysis 1]; Difference in Percentage = 17.5, 95% CI 2-sided [9.3 to 25.5] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in All Participants
Description: DOR was defined as the time from first documented evidence of a confirmed Complete Response (CR) or Partial Response (PR) until progressive disease (PD) or death, whichever occurred first. Per RECIST 1.1 as assessed by BICR, CR was the disappearance of all target lesions and PR was ≥30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. PD was defined as ≥20% increase in the SOD of target lesions according to RECIST 1.1. In addition to the relative increase of 20%, the SOD must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. DOR for participants who had not progressed or died at the time of analysis was censored at the date of the last tumor assessment. DOR was estimated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to 49.5 months
Population: The analysis population included all randomized participants who experienced a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 405 | 331
Months | 8.0 [7.0 to 9.7] | 5.7 [5.5 to 6.9]

11. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1
Description: as for outcome 10
Time Frame: Up to 49.5 months
Population: The analysis population included randomized participants, with a PD-L1 CPS ≥1, who experienced a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 322 | 263
Months | 8.3 [7.0 to 10.9] | 5.6 [5.4 to 6.9]

12. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10
Description: as for outcome 10
Time Frame: Up to 49.5 months
Population: The analysis population included randomized participants, with a PD-L1 CPS ≥10, who experienced a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 169 | 117
Months | 10.9 [8.0 to 13.8] | 5.8 [5.3 to 7.0]

13. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence, in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with at least one AE is presented.
Time Frame: Up to 36.7 months
Population: The analysis population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 785 | 787
Participants | 776 | 771

14. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due To an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to 33.7 months
Population: The analysis population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen)
Number analyzed (Participants) | 785 | 787
Participants | 257 | 204

ADVERSE EVENTS:
Time Frame: Up to 45.9 months
Description: All-cause mortality=all randomized participants and adverse events (AE)=all participants who received ≥1 dose of treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression, malignant neoplasm progression, and disease progression not related to treatment were excluded.
Groups:
- Pembrolizumab Second Course: Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (approximately 2 years) or achieved a complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule of 200 mg IV on Day 1 Q3W for up to 17 cycles (up to approximately 1 year).
Arm/Group | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) | Placebo + Chemotherapy (FP or CAPOX Regimen) | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 601/790 | 666/789 | 2/5
Serious Adverse Events (participants affected / at risk) | 355/785 | 316/787 | 0/5
Other Adverse Events (participants affected / at risk) | 755/785 | 751/787 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) (N=785) | Placebo + Chemotherapy (FP or CAPOX Regimen) (N=787) | Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 8 (10) | 8 (10) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 7 (7) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 5 (5) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 12 (12) | 9 (9) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Ascites (Gastrointestinal disorders) | 5 (6) | 9 (11) | 0 (0)
Colitis (Gastrointestinal disorders) | 16 (16) | 4 (5) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 31 (34) | 25 (26) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 8 (8) | 15 (15) | 0 (0)
Enteritis (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 5 (5) | 7 (7) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (12) | 8 (12) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (3) | 2 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 7 (9) | 5 (6) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 8 (8) | 6 (6) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (14) | 11 (12) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 3 (3) | 9 (9) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Terminal ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (9) | 8 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (20) | 23 (24) | 0 (0)
Asthenia (General disorders) | 4 (4) | 5 (5) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 11 (11) | 4 (4) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 6 (6) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (3) | 0 (0)
Mucosal inflammation (General disorders) | 3 (3) | 5 (5) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 12 (16) | 9 (14) | 0 (0)
Sudden death (General disorders) | 4 (4) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 4 (4) | 2 (3) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (11) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Vanishing bile duct syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 3 (3) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 4 (4) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 3 (3) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lymph node abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 30 (30) | 14 (14) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 7 (8) | 0 (0)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 5 (5) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea manuum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
False positive investigation result (Investigations) | 0 (0) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 7 (7) | 7 (9) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 10 (11) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8) | 6 (7) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 4 (7) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (4) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraneoplastic encephalomyelitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (3) | 0 (0)
Stent malfunction (Product Issues) | 0 (0) | 1 (2) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 12 (13) | 11 (11) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 6 (6) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 3 (3) | 0 (0)
Jugular vein embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy (FP or CAPOX Regimen) (N=785) | Placebo + Chemotherapy (FP or CAPOX Regimen) (N=787) | Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 323 (503) | 284 (412) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 47 (75) | 42 (79) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 28 (37) | 15 (24) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 146 (306) | 141 (294) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 93 (144) | 83 (138) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 20 (23) | 15 (16) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 44 (45) | 13 (15) | 0 (0)
Hypothyroidism (Endocrine disorders) | 120 (134) | 34 (40) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 39 (43) | 40 (42) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 128 (163) | 109 (135) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 59 (68) | 62 (68) | 0 (0)
Constipation (Gastrointestinal disorders) | 169 (207) | 161 (209) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 255 (439) | 238 (357) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 47 (51) | 39 (45) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 47 (49) | 34 (38) | 0 (0)
Nausea (Gastrointestinal disorders) | 359 (620) | 359 (612) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 56 (72) | 48 (53) | 0 (0)
Vomiting (Gastrointestinal disorders) | 251 (418) | 192 (311) | 1 (1)
Asthenia (General disorders) | 125 (196) | 119 (164) | 3 (3)
Fatigue (General disorders) | 193 (252) | 191 (262) | 0 (0)
Mucosal inflammation (General disorders) | 49 (64) | 38 (50) | 0 (0)
Oedema peripheral (General disorders) | 59 (72) | 53 (59) | 0 (0)
Pyrexia (General disorders) | 83 (129) | 51 (63) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 7 (12) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (13) | 12 (12) | 1 (1)
Alanine aminotransferase increased (Investigations) | 130 (172) | 96 (122) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 181 (279) | 137 (188) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 81 (102) | 68 (79) | 0 (0)
Blood bilirubin increased (Investigations) | 105 (186) | 71 (120) | 0 (0)
Blood creatinine increased (Investigations) | 47 (62) | 40 (44) | 0 (0)
Neutrophil count decreased (Investigations) | 197 (537) | 174 (498) | 0 (0)
Platelet count decreased (Investigations) | 206 (415) | 187 (314) | 0 (0)
Weight decreased (Investigations) | 156 (170) | 145 (159) | 1 (1)
White blood cell count decreased (Investigations) | 106 (320) | 92 (282) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 225 (299) | 216 (292) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 63 (105) | 41 (52) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 147 (210) | 105 (145) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 48 (71) | 45 (51) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 116 (162) | 84 (113) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 54 (67) | 39 (48) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 72 (88) | 55 (66) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 50 (52) | 45 (45) | 0 (0)
Dizziness (Nervous system disorders) | 50 (56) | 37 (42) | 0 (0)
Dysgeusia (Nervous system disorders) | 48 (55) | 37 (44) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 157 (215) | 175 (231) | 0 (0)
Paraesthesia (Nervous system disorders) | 47 (74) | 32 (61) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 139 (189) | 136 (184) | 0 (0)
Insomnia (Psychiatric disorders) | 43 (47) | 52 (55) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (44) | 30 (32) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 195 (227) | 171 (187) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 65 (90) | 21 (30) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 72 (99) | 39 (44) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03675737/Prot_SAP_000.pdf